CLINICAL TRIAL: NCT01801189
Title: A Randomized Placebo-Controlled Study of Whether Pre-operative Pregabalin 300 mg Will Improve Pain Control in Patients Undergoing Laparoscopic Roux-en-Y Gastric Bypass (Bariatric Surgery)
Brief Title: Preoperative Pain Control in Gastric Bypass Surgery Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Legacy Health System (Other)
Responsible Party: Principal Investigator, Valerie Halpin, Principal Investigator, Legacy Health System
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: H001
Record Dates: First submitted 2013-02-05; First posted 2013-02-28 (Estimated); Results first posted 2022-06-06 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Post-operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Pregabalin; Sugars; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pregabalin (Experimental): Single, 300 mg pre-operative oral dose of Pregabalin.
  Interventions: Drug: Pregabalin
- Sugar Pill (Placebo Comparator): Single, placebo pre-operative dose.
  Interventions: Drug: Placebo (for Pregabalin)

INTERVENTIONS:
Drug: Pregabalin — One 300 mg oral dose of Pregabalin given before surgery.
  Other Names: Lyrica
  Arms: Pregabalin
Drug: Placebo (for Pregabalin) — One oral dose of placebo given before surgery.
  Other Names: Sugar pill manufactured to mimic Pregabalin 300 mg tablet
  Arms: Sugar Pill

SUMMARY:
Randomized clinical trial to evaluate whether a single pre-operative dose of Pregabalin will alleviate post-operative pain and decrease post-operative analgesic requirements in morbidly obese patients undergoing laparoscopic gastric bypass surgery.

DETAILED DESCRIPTION:
Pregabalin is a popular adjunct for relieving neuropathic pain in diabetics. There have been multiple studies evaluating its use in pre and post-operative pain control in various surgeries. Post-operative pain control is a challenging problem in bariatric patients due to the high doses of narcotic required, related to the high body mass, and the danger of concomitant respiratory depression. In the obese patient, the goal of postoperative pain management is provision of comfort, early mobilization and improved respiratory function, without causing inadequate pain control, respiratory compromise or increased nausea.

Methods: A Randomized Controlled Trial, whereby patients undergoing Laparoscopic Roux-en-Y gastric bypass will be administered a single pre-operative dose of Pregabalin or a placebo. We plan to follow their immediate post-operative course in the hospital, with regard to the following primary endpoints:

* Post-operative analgesic requirements
* Post-operative pain scale (rated 0-10)
* Episodes of vomiting
* Post-operative antiemetic requirement
* Length of stay

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing laparoscopic Roux-en-Y gastric bypass surgery.

Exclusion Criteria:

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2013-02; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Halpin, MD, Principal Investigator — Legacy Health System
Locations (1):
- Legacy Good Samaritan Medical Center, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pregabalin | Sugar Pill
Started | 28 | 33
Completed | 28 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin | Sugar Pill | Total
Number analyzed (Participants) | 28 | 33 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.89 (9.77) | 50.74 (13.66) | 49.91 (12.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 26 | 46
  Male | 8 | 7 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Pain Medication Requirements
Time Frame: Morphine milligram equivalent opioid requirements on post op days zero, 1, and 2.
Measure: Mean (Standard Deviation); unit: MME
Arm/Group | Pregabalin | Sugar Pill
Number analyzed (Participants) | 28 | 33
MME
  POD 0 | 13.76 (11.61) | 17.32 (9.15)
  POD 1 | 40.89 (28.71) | 46.63 (30.67)
  POD 2 | 33.62 (27.6) | 29.74 (26.08)
Statistical Analysis 1: Comparison: Pregabalin vs Sugar Pill; Test type: Superiority; p = 0.10, t-test, 1 sided — Threshold for significance was P <0.05
Statistical Analysis 2: Comparison: Pregabalin vs Sugar Pill; POD 1; Test type: Superiority; p = .23, t-test, 1 sided — Threshold for significance <0.05
Statistical Analysis 3: Comparison: Pregabalin vs Sugar Pill; POD 2; Test type: Superiority; p = .31, t-test, 1 sided — Threshold for significance <0.05

2. Secondary Outcome: Length of Stay
Description: Length of stay in days after surgical procedure
Time Frame: Days in hospital following surgical procedure, up to 5 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Pregabalin | Sugar Pill
Number analyzed (Participants) | 28 | 33
Days | 2.19 (0.47) | 2.24 (0.6)

ADVERSE EVENTS:
Arm/Group | Pregabalin | Sugar Pill
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/33
Other Adverse Events (participants affected / at risk) | 0/28 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No